CLINICAL TRIAL: NCT02089906
Title: Health Status of Chinese Elderly
Brief Title: Health and Nutrition Status of Chinese Elderly
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: BL22
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Malnutrition; Sarcopenia
MeSH Terms: conditions — Malnutrition; Sarcopenia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chinese Elderly: multi-center cross-sectional study

SUMMARY:
This study is aiming to understand the prevalence and risk factors related to malnutrition and sarcopenia in Chinese elderly.

DETAILED DESCRIPTION:
The study objective is to understand the prevalence of malnutrition and sarcopenia in Chinese elderly with the cut-off points from the normal range of muscle mass and function in Chinese adults; to understand the risk factors related to malnutrition and sarcopenia in Chinese elderly; to set up a screening tool on malnutrition and sarcopenia risks in Chinese elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Chinese ages >= 60 years.
2. Subject lives in the community for more than 12 months.
3. Subject has voluntarily signed and dated an informed consent form, approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) prior to any participation in the study.

Exclusion Criteria:

1. Subject who did/does heavy manual labor
2. Subject who was a professional or semi-professional athlete or game player
3. Subject who has physical disabilities such as loss of hand or foot or limbs or any other physical disability which may affect the muscle mass by the opinion of the study physician.
4. Subject has an implanted electronic device or orthopedic metal implantations, such as pacemaker, cardiac defibrillator, subcutaneous injection pump, or metal hip, metal knee joint, metal fracture internal fixation, etc.
5. Subject who has active hyperthyroidism or hypothyroidism and needs medication treatment as by self-report.
6. Subject who has severe heart dysfunction or renal dysfunction with significant sodium water retention or edema by the opinion of study physicians.
7. Subject who takes hormones except for external application of glucocorticoids.
8. Subject who takes diuretics except for using a stable dose for at least 3 weeks as a part of hypertension treatment.
9. Subject who has later stage of malignancies with cachexia by the opinion of study physicians.
10. Subject has any other disease or situation who should not to participate in the study by the opinion of study physicians.
11. Subject had hand/wrist or foot/leg surgery/injury within the past 3 months and the surgery/injury may affect the hand grip or gait speed test by study physician's opinion.
12. Subject is too frail by study physician's opinion
13. Subject is drug addicted or alcohol addicted
14. Subject is participating in other clinical trials which are not approved by AN

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Multi-center cross-sectional study of community dwelling chinese
Sampling Method: Non-Probability Sample
Enrollment: 2834 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Total skeletal muscle mass | Test Visit 1 (~ Day 7)
  bioelectric impedance absorptiometry (BIA)

SECONDARY OUTCOMES:
Total skeletal muscle mass | Test Visit 2 (~ Day 17)
  Dual X-ray Absorptiometry (DXA)
Total body fat | Test Visit 1 (~Day 7) and Test Visit 2 (~ Day 17)
Hand grip strength | Test Visit 1 (~ Day 7)
Gait speed | Test Visit 1 (~ Day 7)
Total body fat free mass | Test Visit 1 (~ Day 7) and Test Visit 2 (~ Day 17)

CONTACTS AND LOCATIONS:
Overall Officials: Xianfeng Zhao, MD, PhD, Study Chair — Abbott Nutrition China
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Shanghai 6th People's Hospital, Shanghai